CLINICAL TRIAL: NCT02131129
Title: Cortical Activation and Cognitive Performance During Repetitive Transcranial Magnetic Stimulation in First-Episode Psychosis: A Pilot Study
Brief Title: rTMS in First Episode Psychosis
Acronym: EmeraldThunder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Neuronetics (Other)
Responsible Party: Principal Investigator, Michael Francis, Psychiatrist, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1401416429
Record Dates: First submitted 2014-05-02; First posted 2014-05-06 (Estimated); Results first posted 2019-01-29 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-03

CONDITIONS: Schizophrenia; Schizophreniform Disorder; Schizoaffective Disorder
Keywords: schizophrenia; schizophreniform disorder; schizoaffective disorder; first episode; psychosis; cognition
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rTMS (Experimental): The stimulation sites will be the left and right DLPFC, defined as 5 cm anterior to the scalp positions at which the MTs were determined. Treatments will be delivered within the following stimulation parameters: 110% of MT, 20 Hz, 30 trains, 1.0 second per train, 20 pulses per train, inter-train interval of 30 seconds (600 pulses/hemisphere, for a total of 1200 pulses/session/day).
  Interventions: Device: rTMS
- Sham (Sham Comparator): The stimulation sites will be the left and right DLPFC, defined as 5 cm anterior to the scalp positions at which the MTs were determined. Treatments will be delivered within the following stimulation parameters: 110% of MT, 20 Hz, 30 trains, 1.0 second per train, 20 pulses per train, inter-train interval of 30 seconds (600 pulses/hemisphere, for a total of 1200 pulses/session/day).
  Interventions: Device: Sham Comparator

INTERVENTIONS:
Device: rTMS — The stimulation sites will be the left and right DLPFC, defined as 5 cm anterior to the scalp positions at which the MTs were determined. Treatments will be delivered within the following stimulation parameters: 110% of MT, 20 Hz, 30 trains, 1.0 second per train, 20 pulses per train, inter-train interval of 30 seconds (600 pulses/hemisphere, for a total of 1200 pulses/session/day).
  Ten sessions over a two week duration
  Other Names: NeuroStar
  Arms: rTMS
Device: Sham Comparator — The stimulation sites will be the left and right DLPFC, defined as 5 cm anterior to the scalp positions at which the MTs were determined. Treatments will be delivered within the following stimulation parameters: 110% of MT, 20 Hz, 30 trains, 1.0 second per train, 20 pulses per train, inter-train interval of 30 seconds (600 pulses/hemisphere, for a total of 1200 pulses/session/day).
  Ten sessions over a two week duration
  Other Names: NeuroStar
  Arms: Sham

SUMMARY:
This study proposes to examine the application of rTMS for the treatment of cognitive dysfunction in FEP. This is an important population for study because if effective, rTMS may represent a preventative treatment for the development of social and vocational impairment that is associated with cognitive dysfunction in schizophrenia. This study will also seek to refine the understanding of the brain circuitry that mediates the potential pro-cognitive effects of rTMS through the use of functional magnetic resonance imaging (fMRI) at baseline and following the course of rTMS administration.

DETAILED DESCRIPTION:
Schizophrenia is a chronic and disabling illness that typically begins in the late teen and early adult years.1 This illness is associated with significant impairments in areas such as independent living, social functioning, and vocational functioning.2 Indeed, only 10% of people with schizophrenia are employed, translating into annual lost wages of nearly 15 billion dollars.3,4 Schizophrenia also represents an important societal burden as this illness has been estimated to cost over 40 billion dollars each year in the United States alone.5

Repetitive transcranial magnetic stimulation (rTMS) is a novel treatment for neuropsychiatric illness. A non-invasive intervention, rTMS utilizes the application of a repetitively pulsed magnetic field over the scalp to induce an electric field within a discrete area of the cerebral cortex. This electric field results in altered ion flow across the neuronal cellular membrane and ultimately changes in neuronal polarization. The end result is altered neuronal activity in the area of the cerebral cortex where the rTMS is applied.12 rTMS is a safe and well-tolerated intervention that received FDA approval for treatment refractory major depressive disorder in 2008 and has since become commonly used in clinical practice.13

This study proposes to examine the application of rTMS for the treatment of cognitive dysfunction in FEP. This is an important population for study because if effective, rTMS may represent a preventative treatment for the development of social and vocational impairment that is associated with cognitive dysfunction in schizophrenia. This study will also seek to refine the understanding of the brain circuitry that mediates the potential pro-cognitive effects of rTMS through the use of functional magnetic resonance imaging (fMRI) at baseline and following the course of rTMS administration.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years of age at study entry
* Male or female
* DSM IV-TR Diagnosis of schizophrenia, schizophreniform disorder, or schizoaffective disorder as confirmed by Structured Clinical Interview for DSM-IV-TR (SCID)44
* Subjects in their first-episode of psychosis, defined as the onset of clinically significant psychotic symptoms within the past five years as determined by first medical record documentation of these conditions
* BACS composite t-score of 40 or less at baseline assessment
* Clinical stability as defined by:

  * CGI-S score of less than or equal to 4 (moderately ill) at randomization AND
  * Subjects must not have experienced an exacerbation of their illness within 4 weeks prior to randomization, leading to an intensification of psychiatric care in the opinion of the investigator. Examples of intensification of care include, but are not limited to: inpatient hospitalization, day/partial hospitalization, outpatient crisis management, or psychiatric treatment in an emergency room AND
  * Antipsychotic treatment stability for at least 4 weeks prior to randomization (no change in antipsychotic dosing or addition of any new antipsychotic medication).
* Able to give informed consent
* Subjects must be willing and able to adhere to study schedule
* Outpatient or Inpatient treatment status
* Female subjects of childbearing potential must test negative for pregnancy at screening and baseline visit

Exclusion Criteria:

* Life-time history of a seizure, excluding febrile seizures and those induced by substance withdrawal
* Metallic objects planted in or near the head, including implanted pacemaker, medication pump, vagal stimulator, deep brain stimulator, TENS unit, ventriculoperitoneal shunt, or cochlear implants
* First degree relative (that is, biological father, mother, brother, sister, or child) with idiopathic epilepsy or other seizure disorder
* History of significant neurological illness (including stroke, CNS infection with persistent neurologic deficit, or other event deemed significant by PI)
* History of head trauma as defined by a loss of consciousness or a post-concussive syndrome deemed significant by PI
* Pregnancy or breast feeding
* Known IQ < 70 based on medical history
* Current DSM-IV-TR diagnosis of alcohol or drug dependence (excluding nicotine or caffeine)
* Subjects with current acute, serious, or unstable medical conditions, including, but not limited to: inadequately controlled diabetes, asthma, COPD, severe hypertriglyceridemia, recent cerebrovascular accidents, acute systemic infection or immunologic disease, unstable cardiovascular disorders, malnutrition, or hepatic, renal gastroenterological, respiratory, endocrine, neurologic, hematologic, or infectious diseases based on medical history or physical examination.
* Subjects with contraindications to MRI or otherwise unable to tolerate MRI procedure
* Subjects considered a high risk for suicidal acts - active suicidal ideation as determined by clinical interview OR any suicide attempt in 90 days prior to screening
* Subjects who have participated in a clinical trial with any pharmacological treatment intervention for which they received study-related medication in the 4 weeks prior to randomization
* Subjects who require concomitant treatment with prohibited medication, as specified in Attachment 2
* Subjects with a history of electroconvulsive therapy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04-30 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - IU Center for NeuroImaging, Indianapolis, Indiana
  - Prevention and Recovery Center for Early Psychosis, Indianapolis, Indiana

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period for the study was from 04/2014-09/2016. Recruitment took place at the Prevention and Recovery Center for Early Psychosis, an Eskenazi Health - Midtown Mental Health Clinic and at local community mental health centers in the Indianapolis area.
Groups:
- rTMS: The stimulation sites will be the left and right DLPFC, defined as 5 cm anterior to the scalp positions at which the MTs were determined. Treatments will be delivered within the following stimulation parameters: 110% of MT, 20 Hz, 30 trains, 1.0 second per train, 20 pulses per train, inter-train interval of 30 seconds (600 pulses/hemisphere, for a total of 1200 pulses/session/day).
  rTMS: The stimulation sites will be the left and right DLPFC, defined as 5 cm anterior to the scalp positions at which the MTs were determined. Treatments will be delivered within the following stimulation parameters: 110% of MT, 20 Hz, 30 trains, 1.0 second per train, 20 pulses per train, inter-train interval of 30 seconds (600 pulses/hemisphere, for a total of 1200 pulses/session/day).
  Ten sessions over a two week duration
- Sham: The stimulation sites will be the left and right DLPFC, defined as 5 cm anterior to the scalp positions at which the MTs were determined. Treatments will be delivered within the following stimulation parameters: 110% of MT, 20 Hz, 30 trains, 1.0 second per train, 20 pulses per train, inter-train interval of 30 seconds (600 pulses/hemisphere, for a total of 1200 pulses/session/day).
  Sham Comparator: The stimulation sites will be the left and right DLPFC, defined as 5 cm anterior to the scalp positions at which the MTs were determined. Treatments will be delivered within the following stimulation parameters: 110% of MT, 20 Hz, 30 trains, 1.0 second per train, 20 pulses per train, inter-train interval of 30 seconds (600 pulses/hemisphere, for a total of 1200 pulses/session/day).
  Ten sessions over a two week duration
Period: Overall Study
Arm/Group | rTMS | Sham
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rTMS | Sham | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23.4 (3.1) | 22.3 (2.0) | 22.8 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 7 | 8 | 15
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Performance
Description: rTMS effectiveness in improving cognitive performance as measured by the Brief Assessment of Cognition in Schizophrenia (BACS) composite score. The BACS is a battery specifically designed to measure treatment-related changes in cognition, and has alternate forms, thus minimizing practice effects. The battery includes brief assessments of executive functions, verbal fluency, attention, verbal memory, working memory and motor speed, and generates a composite score that is calculated by summing t-scores derived by comparisons with a normative sample of 404 healthy controls. The six brief assessments' t-scores, are summed, and averaged to provide a composite t-score. The composite score min and max are between -43 and 100. A higher score indicating better cognitive performance. The composite score is reported as a change score relative to baseline for both.
Time Frame: For within-group comparisons, scores at V13 (day 15) and V14 (follow-up two weeks after V13) were compared to baseline
Measure: Least Squares Mean (Standard Error); unit: BACS Composite Score
Arm/Group | rTMS | Sham
Number analyzed (Participants) | 9 | 10
BACS Composite Score
  BACS Composite Score at V13 | 2.22 (2.86) | -0.50 (2.72)
  BACS Composite Score at V14 | 6.11 (2.86) | -3.70 (2.72)

2. Primary Outcome: Cortical Activation
Description: effects of rTMS on cortical activation using fMRI during working memory and episodic memory tasks
Time Frame: Change from Baseline (day 1) to Visit 13 (day 15)
Measure: Mean (Standard Deviation); unit: Bold signal change
Arm/Group | rTMS | Sham
Number analyzed (Participants) | 9 | 10
Bold signal change | 0.099872925 (0.196355152) | 0.115569747 (0.297909567)

3. Secondary Outcome: Cognitive Performance
Description: rTMS effectiveness in improving cognitive performance was assessed by the Trail Making Test-Part B change score and performance on the Trail Making Test-Part B. The Trail Making Test-Part B is a measure of visual attention and task switching. The task requires a subject to 'connect-the-dots' of 25 consecutive targets on a sheet of paper. In Part B version the subject alternates between numbers and letters (1, A, 2, B, etc.) The goal of the test is for the subject is to finish part B as quickly as possible, the time taken to complete the test is used as the primary performance metric.
Time Frame: 14 days
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | rTMS | Sham
Number analyzed (Participants) | 9 | 10
seconds | 107.8 (24.4) | 83.3 (29.0)

4. Secondary Outcome: Cognitive Performance
Description: rTMS effectiveness in improving cognitive performance as measured by the Brief Assessment of Cognition in Schizophrenia (BACS) composite score. The BACS is a battery specifically designed to measure treatment-related changes in cognition by utilizing 6 tasks, and has alternate forms, thus minimizing practice effects. Each task generates a raw score (with a higher score indicating better performance): verbal memory 0-75; digit sequencing 0-28; token motor task 0-100; semantic&letter fluency 0-148; symbol coding 0-110; and tower of London 0-22. The raw scores are used to generate a composite score that is calculated by summing t-scores derived by comparisons with a normative sample of 404 healthy controls. The six brief assessments' t-scores, are summed, and averaged to provide a composite t-score. The composite score min and max are between -43 and 100. A higher score indicating better cognitive performance.
Time Frame: 14 days
Measure: Least Squares Mean (Standard Error); unit: BACS Sub-scale Scores
Arm/Group | rTMS | Sham
Number analyzed (Participants) | 9 | 10
BACS Sub-scale Scores
  Verbal Memory | 0.78 (2.53) | -6.30 (2.40)
  Digit Sequencing | 1.11 (2.69) | 1.40 (2.55)
  Token Motor Total | 11.00 (4.99) | 3.80 (4.74)
  Semantic & Letter Fluency | 3.33 (2.90) | -7.00 (2.75)
  Symbol Coding | 4.78 (2.89) | -3.80 (2.74)
  Tower of London | 0.44 (5.13) | -0.90 (4.87)

5. Secondary Outcome: Symptoms
Description: rTMS effectiveness in general symptomatology assessed by the Positive and Negative Syndrome Scale (PANSS). The PANSS is a semi-structured interview, containing 30 items that assess symptoms of psychotic disorders including positive, negative, and general psychopathology symptoms. Positive symptoms are rated on 7 items, negative symptoms are rated on 7 items, and general psychopathology on 16 items. Scores for each item range from 1=absent to 7=extreme. Positive, negative, and general psychopathology symptoms can each respectively render total scores. Positive total scores ranging from 7-49, negative total scores ranging from 7-49, and general psychopathology scores ranging from 16-112. When all items are summed together a total score is generated. Total scores for all items range from 30-210, a lower score reflecting fewer symptoms.
Time Frame: For within-group comparisons, scores at V13 (day 15) and V14 (follow-up two weeks after V13) were compared to baseline
Measure: Least Squares Mean (Standard Error); unit: Change Scores Relative to Baseline
Arm/Group | rTMS | Sham
Number analyzed (Participants) | 9 | 10
Change Scores Relative to Baseline
  V13 PANSS Total Score | -0.89 (3.12) | 5.60 (2.96)
  V14 PANSS Total Score | -1.11 (3.12) | 6.80 (2.96)
  V13 PANSS Total Negative Score | 1.33 (1.90) | 2.00 (1.80)
  V14 PANSS Total Negative Score | -0.11 (1.90) | 2.00 (1.80)
  V13 PANSS Total Positive Score | -1.44 (1.17) | 1.60 (1.11)
  V14 PANSS Total Positive Score | -0.78 (1.17) | 2.50 (1.11)

6. Secondary Outcome: Negative Symptoms
Description: rTMS effectiveness in reducing negative symptoms as measured by the negative symptom assessment scale (NSA-16). The NSA-16 is used to help clinicians rate behaviors (not psychopathology) commonly associated with negative symptoms of schizophrenia. The scale rates subjects on 16 "anchors," is a semi-structured, clinical interview, and each item is rated from 1 to 6. The total score is the sum of the 16 specific items and ranges from 16 to 96; a higher score indicates greater severity of illness. In addition, there is a global rating that represents the overall assessment of a subject's negative symptoms. The rating should not be an average of any particular behavior, but a gestalt of everything observed in the interview.
Time Frame: Assessed at Baseline (day 0), Midpoint (day 8), and Endpoint (day 15)
Measure: Mean (Standard Deviation); unit: NSA-16 Scores
Arm/Group | rTMS | Sham
Number analyzed (Participants) | 9 | 10
NSA-16 Scores
  NSA-16 Total Baseline Scores | 40.67 (12.49) | 44.80 (11.58)
  NSA-16 Total Midpoint Scores | 46.44 (16.45) | 46.40 (12.86)
  NSA-16 Total Endpoint Scores | 42.22 (14.93) | 46.90 (17.04)

ADVERSE EVENTS:
Arm/Group | rTMS | Sham
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 4/10 | 3/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rTMS (N=10) | Sham (N=10)
Right Earache (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (4)
Gum Sensation (Nervous system disorders) | 0 (0) | 1 (1)
Muscle Twitch (post treatment) (Nervous system disorders) | 0 (0) | 1 (1)
Application Site Discomfort (Nervous system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No